CLINICAL TRIAL: NCT02781012
Title: Project Survival-Prospective Biomarker Discovery to Transform Diagnosis and Treatment for Patients With Pancreatic Diseases and Cancer
Brief Title: Project Survival-Prospective Biomarker Discovery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pancreatic Cancer Research Team (Other)
Collaborators: BPGbio (Industry)
Responsible Party: Sponsor
Other Study IDs: PCRT 15-001
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer; Pancreatitis; Pancreatic Adenocarcinoma; Metastatic Pancreatic Cancer
Keywords: Pancreatic Disease; Pancreas; Borderline Resectable; Pancreatic Cancer; Pancreatitis; Family history of pancreatic cancer; Healthy; Healthy at risk
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood (serum, plasma, buffy coat), saliva, urine, and pancreatic tissue designated as surgical waste by site's treating pathologist.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy: Healthy volunteers without any known pancreatic disease
- Healthy At-Risk: Healthy volunteers with no known benign or malignant pancreatic disease, AND with one first-degree relative with pancreatic cancer, OR two second-degree relatives with pancreatic cancer. These subjects also include those who have undergone surgery for suspected pancreatic cancer, and who are found to have a non-pancreatic cancer pathology upon final local site or central pathology review.
- Pancreatitis: Subjects diagnosed with acute or chronic pancreatitis
- Early Stage/Borderline/Locally Advanced: Subjects diagnosed with early stage pancreatic cancer who undergo surgery as standard of care therapy with or without preoperative (neoadjuvant) chemotherapy and/or radiation therapy; subjects diagnosed with borderline pancreatic cancer, or subjects diagnosed with locally advanced pancreatic cancer.
- Metastatic: Subjects diagnosed with metastatic pancreatic cancer and treated with any standard of care therapy/therapies.

SUMMARY:
This sample-collection study is open to participants in several categories: healthy volunteers (with or without a family history of pancreatic cancer) and individuals diagnosed with pancreatitis or any stage of pancreatic cancer. All participants will submit urine, saliva and blood samples; pancreatitis and pancreatic cancer patients will also submit tissue samples if biopsy/ies or surgery is part of the care being provided by their doctor. In partnership with Berg Health, LLC, biomarkers will be investigated for potential use in early detection of pancreatic cancer, to determine prognosis of patients, and to find the most appropriate treatments for patients.

DETAILED DESCRIPTION:
The Primary Objective of this study is to identify and validate biomarkers that can be used for early detection and selection of personalized treatment of pancreatic diseases, including adenocarcinoma and pancreatitis. A maximum of 600 subjects will be enrolled in this study, including healthy volunteers, subjects with acute and chronic pancreatitis, family members at risk for pancreatic cancer (as defined below), and subjects with all stages of pancreatic adenocarcinoma who will contribute samples annotated with longitudinal clinical data. Biomarkers will be investigated for potential as Theranostic, Prognostic, Diagnostic and Therapeutic indicators among subjects with pancreatitis and pancreatic cancer.

Examples of eligible participants include:

* Healthy volunteers without any known pancreatic disease (50 subjects)
* Healthy volunteers with no known benign or malignant pancreatic disease, AND with one first-degree relative with pancreatic cancer, OR two second-degree relatives with pancreatic cancer. These subjects also include those who have undergone surgery for suspected pancreatic cancer, and who are found to have a non-pancreatic cancer pathology upon final local site or central pathology review. (100 subjects).
* Subjects diagnosed acute or chronic pancreatitis (50 subjects).
* Subjects diagnosed with early stage pancreatic cancer who undergo surgery as standard of care therapy with or without preoperative (neoadjuvant) chemotherapy and/or radiation therapy; subjects diagnosed with borderline pancreatic cancer, or subjects diagnosed with locally advanced pancreatic cancer (200 subjects). Enrollment of treatment naïve subjects with early stage pancreatic cancer is preferred.
* Subjects diagnosed with metastatic pancreatic cancer and treated with any standard of care therapies, such as gemcitabine/Abraxane or FOLFIRINOX as front-line treatment with or without associated radiation treatment (200 subjects). Enrollment of treatment naïve subjects with metastatic pancreatic cancer is preferred.

Consented and enrolled subjects will be asked to participate in this study in the following ways:

* Subjects will be asked to contribute blood (serum, buffy coat, and plasma), urine, and saliva after enrollment, and at clinically-significant timepoints throughout their treatment as indicated by their disease state.
* Subjects undergoing surgery for pancreatic disease will also be asked to donate diseased and adjacent non-diseased pancreatic tissue, defined as "excess" tissue from diagnostic or therapeutic biopsy or surgical procedures that is no longer required for standard of care purposes.
* Examples of "excess" tissue after a standard of care surgical procedures include any/all biopsies or resections performed and may include non-diseased pancreatic tissue and pancreatic tumor tissue.
* These collection procedures will not alter or prolong the conduct of standard of care surgical procedures.

Subsequent liquid non-tissue samples will be collected from all subjects at the following clinically-relevant time points related to standard of care treatment for pancreatic disease:

* Before, at the time of, and/or after surgery to remove a pancreatic tumor or inflammatory mass;
* before and after chemotherapy and/or radiation for cancer;
* upon local, regional, or distant progression of cancer;
* resolution of the disease process.

Blood (serum, plasma, and buffy coat), urine and saliva will not be collected more than six (6) times in a 12 month period per subject.

Samples will be collected until the subject withdraws or the study has completed enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is over 18 years of age and has been evaluated at a participating Pancreatic Cancer Research Team (PCRT) study site, AND
2. Subject has been recently diagnosed with pancreatic cancer (any stage) OR
3. Subject has been recently (within 12 months) diagnosed with acute or chronic pancreatitis OR
4. A healthy individual, with no known pancreatic disease (cancerous or otherwise), AND with one first-degree relative with pancreatic cancer, OR two second-degree relatives with pancreatic cancer OR one who has undergone surgery for suspected pancreatic cancer, and who is found to have a non-pancreatic cancer pathology upon final local site or central pathology review, OR
5. A healthy individual with no known benign or malignant pancreatic disease, and no family history of pancreatic cancer.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Subject is < 18 years old.
* Subject has been diagnosed with a primary cancer other than pancreas in the past 5 years, and is currently receiving treatment for this cancer.
* Subject is a pregnant or lactating female;
* Subject is not willing or is unable to give informed consent to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants in several categories:
  * Healthy Volunteers,
  * Healthy At-Risk Volunteers (whose immediate or extended family member(s) were diagnosed with Pancreatic Cancer),
  * Patients with a suspected malignant tumor in pancreas who require surgery,
  * Pancreatitis Patients (both Acute and Chronic), and
  * Patients with all stages of Pancreatic Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2016-03; Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Berg's Interrogative Biology® Platform | Sample analysis will occur throughout enrollment period (5 years), and outcomes will be assessed at end of enrollment period.
  Tissue and fluid samples will be analyzed using Berg's Interrogative Biology® Platform, which uses biomolecular analyses paired with artificial intelligence to identify and validate biomarkers that can be used for early detection of pancreatic diseases, including pancreatic cancer, and to determine the prognosis of patients, and best therapeutic treatment for specific patients.

CONTACTS AND LOCATIONS:
Overall Officials: A. James Moser, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard University; Tomislav Dragovich, MD, Principal Investigator — Banner Health - MD Anderson Cancer Center
Locations (6):
- United States (6):
  - Banner Health - MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mercy Health - St. Mary's, Grand Rapids, Michigan
  - Virginia Piper Cancer Institute - Allina Health, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project Survival Patient Information Webpage — https://pcrt.crab.org/ProjectSurvival.aspx